CLINICAL TRIAL: NCT00346827
Title: Apomorphine Nasal Powder in the Treatment of Parkinson's Disease "Off" Periods.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Britannia Pharmaceuticals Ltd. (Industry)
Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20102D05
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: 3-week, double-blind, placebo-controlled, 3 × crossover efficacy phase followed by 12 week open label phase, followed by 36 week open continuation phase
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Apomorphine Nasal Powder

SUMMARY:
To determine the safety and tolerability of repeated dosing with Apomorphine Nasal Powder in subjects with Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* 1 year history of Parkinson's Disease; stable PD medications for 4 weeks; at least one documented "off" period per day

Exclusion Criteria:

* hypersensitivity to apomorphine; participation in a clinical trial in the last 12 weeks; pregnant or lactating females

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Weiser, MB, MRCP, Principal Investigator — Swansea Hospital, Swansea, Wales